CLINICAL TRIAL: NCT06577974
Title: Does the Medical Tretament Prior to Stimulation Affect the Fertility Outcome in Cases of Endometriosis Associated Infertiltiy
Brief Title: Role of Medical Treatment in Endometriosis Patients Undergoing ICSI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mariam Ahmed Mohamed Dawoud, Associate professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MD-70-2023
Record Dates: First submitted 2024-08-16; First posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Endometriosis
Keywords: Oocyte yield, fertilisation rate
MeSH Terms: conditions — Endometriosis | interventions — drospirenone and ethinyl estradiol combination; dienogest

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Those treated by COCPs before IVSI (Experimental): Those with endometrisosis who will undergo ICSI after pretreatment with COCPs
  Interventions: Drug: Combined contraceptive pills (Yasmin)
- Those treated by Dionogest before ICSI (Experimental): Patients diagnosed with endometriosis who will undergo ICSI after oreteatment by dienogest
  Interventions: Drug: Combined contraceptive pills (Yasmin)
- Those undergoing ICSI straighaway (No Intervention): patients diagnosed with endometriosis who will undergo ICSI without any medical pretretament

INTERVENTIONS:
Drug: Combined contraceptive pills (Yasmin) — medical pretreatment prior to ICSI
  Other Names: Dienogest (Visanne)
  Arms: Those treated by COCPs before IVSI; Those treated by Dionogest before ICSI

SUMMARY:
The aim of this study to assess the effect of medical treatment prior to stimulation on fertility (ICSI) outcome in cases with endometriosis associated infertility.

DETAILED DESCRIPTION:
Patients complaining of infertility due to endometriosis diagnosed by ultrasound or laparoscopic surgery will be randomly allocated to three groups :

Group A: will receive COCPs for 3-6 months prior to starting IVF / ICSI cycle. Group B: will receive Dienogest for 3-6 months prior to starting IVF / ICSI cycle.

Group C: will be subjected to direct ICSI /IVF cycle. Then all patients will be subjected to ovarian stimulation regimen using GnRH Agonist Down-Regulation Gonadotropin Stimulation-The "Long" Protocol.

During the ovarian stimulation, the woman's response is monitored with serum estradiol levels and vaginal ultrasound examinations. The estradiol level is used to determine the dose of gonadotropins and whether under- or overstimulation occurs. The goal of the ovarian hyperstimulation is to develop at least three mature follicles that are 17 mm in diameter or larger. Once this is achieved, FSH and other medications are discontinued, and a single injection of hcg is given to mature the eggs to allow fertilization.

The hcg administration will also cause ovulation, but this does not occur until 40 hours or later after the injection. Therefore, it is standard that the hcg injection is administered 36 hours before the scheduled egg retrieval such that this will allow adequate maturation of the eggs and yet there would be little risk of ovulation.

Then the process will be continued through oocyte retrieval, oocyte maturation , fertilization by ICSI.

Each group will be followed up to detect the number of oocyte yield, fertilization rate and availability of good quality embryos and then according to the results the effect of medical treatment prior to stimulation will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Presence of Endometrioma on ultrasound.
* History of ovarian cystectomy either open or via laparoscopic surgery.
* Presence of endometriotic foci in the pelvis during laparoscopic surgery.
* Patients coming for the first ICSI / IVF cycle.

Exclusion Criteria:

* Age above 40 years
* Cases with endometrioma on ultrasound more than 3 cm size.
* Prior failed ICSI / IVF.
* Known poor responders or poor ovarian reserve, defined as AFC<5 or AMH < 0.5 .
* Patients with previous uterine surgery.
* Patients diagnosed to have uterine abnormalities

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 129 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Fertilisation rate | 2 weeks from starting induction
  Number of embryos

SECONDARY OUTCOMES:
clinical pregnancy rate | 2 weeks from embryo transfer
  appearance of intrauterine gestational sac

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Taha, Professor, Study Chair — Cairo University
Locations (2):
- Egypt (2):
  - ART unit, Obstetrics and Gynecology Department, Cairo University, Cairo
  - Cairo University/Obstetrics and Gynecology Department/ART Unit, Cairo

IPD SHARING:
Plan to Share IPD: No
Study protocol, excel sheet